CLINICAL TRIAL: NCT06318364
Title: Analysis of the Incidence and Influencing Factors of Postoperative Delirium in the Post-anesthesia Care Unit: A Multicenter, Observational, Matched Case-control Study
Brief Title: Postoperative Delirium in the Post-anesthesia Care Unit
Status: Recruiting | Type: Observational
Sponsor: Qin Zhang (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Qin Zhang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202402016
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Delirium, Postoperative
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients staying in the PACU: Patients staying in the PACU
  Interventions: Other: NO Intervention

INTERVENTIONS:
Other: NO Intervention — NO Intervention

SUMMARY:
This study aims to investigate the incidence of postoperative delirium (POD) in the PACU and analyze its influencing factors, in order to provide theoretical basis for early screening and intervention for high-risk POD population. Blood samples of some study subjects will be collected and analyzed using molecular detection methods to provide a basis and insights into the pathophysiological mechanisms of POD.

DETAILED DESCRIPTION:
Study design type: Multi-center, observational, case-control study based on propensity score matching. The leading unit is Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, and the participating unit is The First Hospital of Harbin Medical University.

Record general clinical information, surgical-anesthesia-related information, recovery indicators, pain status, adverse events in PACU, and occurrences of postoperative delirium of all study subjects meeting the inclusion criteria of this study. Based on the occurrence of postoperative delirium, the subjects will be divided into delirium group and non-delirium group for univariate analysis. Univariate factors with statistical significance will be included in a multiple logistic regression analysis to further identify risk factors for postoperative delirium. Some selected factors can undergo ROC curve analysis to calculate the optimal cutoff value. Due to the limited number of subjects experiencing postoperative delirium, propensity score matching will be used to improve the statistical efficiency for analysis of risk factors for postoperative delirium. Furthermore, for patients with postoperative delirium, a small amount of blood samples will be collected by the researchers for analysis of inflammatory factors and other components.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participating in this study
2. Age ≥18 years old
3. ASA classification I-IV
4. Complete clinical data

Exclusion Criteria:

1. ASA classification V and above
2. History of severe central nervous system diseases, psychiatric disorders, cognitive impairment, intellectual disability, or Mini-Mental State Examination (MMSE) score ≤23
3. Patients with communication barriers
4. Patients with missing clinical data
5. Patients with severe complications during PACU observation requiring reintubation, reoperation, or transfer to the intensive care unit for further treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients entering the PACU and meeting the inclusion criteria of this study
Sampling Method: Probability Sample
Enrollment: 3320 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | 1 Hour
  Mini-Mental State Examination, MMSE

CONTACTS AND LOCATIONS:
Overall Officials: Qin Zhang, Principal Investigator — Tongji Medical College, Huazhong University of Science and Technology
Locations (2):
- China (2):
  - The First Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei